CLINICAL TRIAL: NCT05267067
Title: Comparison Between the Manual Respiratory Exercises and Respiratory Pressure Meter
Brief Title: Impact of Positive End Maximum Voluntary Ventilation and Dyspnea Index in Patients After Valvular Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sahar Ahmed Abdalbary, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Chest physiotherapy
Record Dates: First submitted 2022-02-13; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Respiration Disorders
MeSH Terms: conditions — Respiration Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual respirtory exercises (Active Comparator): Using manual traditional respiratory exercises.
  Interventions: Other: respiratory exercises
- Respiratory exercises with respiratory pressure meter (Active Comparator): Using pressure respiratory meter in exercises.
  Interventions: Other: respiratory exercises

INTERVENTIONS:
Other: respiratory exercises — Manual respiratory exercises versus respiratory exercises with pressure meter

SUMMARY:
Pulmonary mechanics are further disturbed after cardiothoracic surgery that manifests like restrictive pathology, which may persist for weeks to months postoperatively. This experimental aimed to investigate the efficacy of a positive end-expiratory pressure device on maximum expiratory pressure, maximum voluntary ventilation, and dyspnea index in patients who underwent valve surgery.

DETAILED DESCRIPTION:
Thirty male and female adolescent patients who underwent valve surgery aged 12-18 years old, recruited from the national heart institute enrolled in this experimental. They were assigned into two matched groups: Experimental group consisted of 15 patients, received positive end-expiratory pressure (PEEP) with a mouthpiece in addition to routine chest physiotherapy (postural drainage, percussion, vibration, and deep breathing exercises). Control group consisted of 15 patients, received routine chest physiotherapy alone. The program continued for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* underwent valve surgery (repair or replacement) for mitral valve stenosis;
* hemodynamically stable,
* ages ranged from 12 to 18 years old-
* BMI ranges from 18.5 to 24.9
* reduced MEP, MVV and complaining from shortness of breath with exertion.

Exclusion Criteria:

* Patients with previous cardiac surgery
* congenital heart disease
* neurological disorders
* type1 diabetes mellitus
* smoker
* pacemaker implantation
* atrial fibrillation
* utilization of mechanical ventilation longer than 24 hours.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 3 month
  By respiratory pressure meter

CONTACTS AND LOCATIONS:
Overall Officials: Abdallaha Mohamed, MD, Study Chair — Nahda University, Faculty of Physical Therapy
Locations (1):
- Sahar Abdalbary, Cairo, Select State/province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided